CLINICAL TRIAL: NCT04876872
Title: The Effectiveness of Modified Pediatric Early Warning Score and Pediatric Hospitalization Risk Scoring II in Patients Applying to the Pediatric Emergency Unit During Pandemic Period Associated With COVID-19 Disease
Brief Title: Modified Pediatric Early Warning Score and Modified PRISA II During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ahmet Kagan Ozkaya, Karadeniz Technical University, Head of Department of Pediatric Emergency, Karadeniz Technical University
Other Study IDs: KTU-PediEM01
Record Dates: First submitted 2021-05-03; First posted 2021-05-07 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Critical Illness
Keywords: critically ill child; pediatric early warning score; mPEWS; mPRISA II
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients: whole pediatric patients who admitted to the pediatric emergency unit in Farabi Hospital, Trabzon, Turkey
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
One of the most important factors in pediatric emergency units is the correct decision of the patient inpatient or outpatient treatment.

If the disease progresses critically, the decision of hospitalization comes to the fore. However, in this case, it is very important to make the right decision and to determine the situation in a short time.

Children give different physiological responses to diseases according to age group. For this reason, some scoring, which require objective parameters, have been developed in order to predict the critical processes of the patients and to intervene at the right time.

While such scoring is frequently used in adult emergency units, it is understood that studies on this issue are not sufficient in pediatric emergency units.

The purpose of our study; To evaluate the population of children admitted to the pediatric emergency unit with the modified Pediatric Early Warning Scoring (mPEUS) and Pediatric Hospitalization Risk Scoring II (PRISA II), to predict hospitalization and discharge from the emergency service, and to demonstrate the effectiveness of the scoring to identify critically ill children in the correct early period.

DETAILED DESCRIPTION:
Triage is the primary step where the first treatment service of a patient admitted to the emergency unit is initiated.

The purpose of triage in the emergency room is a rapid assessment to determine the order of priority. Emergency service triage systems have been developed mainly to identify the "most urgent" or potentially "critical pediatric" cases and give priority to treatment for these patients.

If the patient's condition is critical in the pediatric emergency unit, the decision for outpatient treatment / hospitalization should be made quickly but in the most correct way. Regardless of the diagnosis, the main problem is; early diagnosis of the critical patient, directing the patient to the appropriate area in the emergency department for acute stabilization, and more importantly, to decide quickly whether the patient will be hospitalized in order to continue the treatment and accelerate the flow of the emergency service. It is known that children who unexpectedly worsen in the hospital environment will have observable features in the period before the seriousness of their condition is understood. It has been emphasized in the studies conducted that ways to understand early whether there is a problem in a child should be investigated. For this reason, some scores that require objective parameters have been developed in order to predict the critical processes of the patients and to intervene at the right time. These scores should be viewed not only as a score, but as a complementary systematic approach used to improve pediatric patient safety and clinical outcomes. mPEUS; These are physiology-based scoring systems developed to identify patients with clinical worsening. Studies have reported that with these scores, the treatment of critical emergency patients can be started without delay. mPEUS has been developed to provide a reproducible assessment of the pediatric patient's condition based on physiological parameters. In addition, the use of these scores in the emergency service and inpatient services ensures continuity in patient evaluation. To date, there are very few data regarding the use of mPEUS in children presenting to the emergency department. Although many mPEUS have been developed and tested, uncertainty remains as to which system or system feature is most beneficial for pediatric patients. Therefore, studies on this subject should be increased. mPEUS is an essential tool for patient safety. The use of mPEUS during the initial evaluation can help prevent poor neurological results, deterioration of the patient's condition, and reduce mortality with rapid intervention. In limited studies conducted in pediatric emergency units, it has been shown that these early warning scores can determine the children who need to be admitted to the Pediatric Intensive Care Unit (PICU). With this scoring, the early hospitalization of the patient in the emergency room can be accurately predicted. Such early warning scoring can be used to shorten patients' hospitalization and waiting times in emergency rooms. The PRISA II system, similar to mPEUS but used only to predict inpatients, has also been developed. This scale includes initial history, physiological parameters, chronic disease status, treatments applied in the emergency department and laboratory values. It is appropriate to use PRISA II to control the severity of the disease. There is not enough data in the literature regarding the efficacy of both mPEUS and PRISA II scoring in the epidemic period associated with COVID-19. With this study, it is aimed to provide efficiency by using these scoring in patients who applied to the pediatric emergency unit during the pandemic period.

ELIGIBILITY:
Inclusion Criteria:

- Pediatric patients aged between 28 days and 18 years, who applied to the Pediatric Emergency Unit

Exclusion Criteria:

* In the follow-up or at the begining, patients who are presenting with cardiorespiratory arrest
* Intubated patients,
* Trauma patients
* Neonatal period (<28 days),
* Patients who leave the hospital at the request of their family before the end of the diagnosis or treatment process
* Patients who do not have permission from their parents at the beginning

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients aged between 28 days and 18 years who applied to the Pediatric Emergency Unit
Sampling Method: Non-Probability Sample
Enrollment: 894 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
modified pediatric early warning score | 1 February - 31 July 2021,
  modified pediatric early warning score for each child during Severe Acute Respiratory Syndrome Causing Coronavirus Disease
mPRISA II | 1 February - 31 July 2021
  mPRISA II score for each child during COVID-19 pandemic
Changes in modified pediatric early warning score over time | 1 February - 31 July 2021
  Changes in modified pediatric early warning score over time will measure. Early warning score will be calculated every three hours and if the score increases, it will be evaluated more frequently, up to 24 hours.

SECONDARY OUTCOMES:
Length of stay in pediatric emergency | 1 February - 31 July 2021
  Length of stay in pediatric emergency
number of children who returned to the emergency service | 1 February - 31 July 2021
  number of children who returned to the emergency service
which service is admitted to | 1 February - 31 July 2021
  pediatric wards
number of children with severe acute respiratory syndrome coronavirus 2 | 1 February - 31 July 2021
  Children diagnosed with COVID-19 (real time PCR positive children)
children who contacted the person with COVID-19 | 1 February - 31 July 2021
  number and status of children who contacted the person with COVID-19
history of COVID-19 in the past | 1 February - 31 July 2021
  number of children who had COVID-19 in the past

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet K Özkaya, MD, phD, Study Director — Karadeniz Technical University Faculty of Medicine; Bihter Şen Şahin, MD, Principal Investigator — Karadeniz Technical University Faculty of Medicine
Locations (1):
- Karadeniz Technical University Faculty of Medicine Farabi Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamberlain JM, Patel KM, Pollack MM. The Pediatric Risk of Hospital Admission score: a second-generation severity-of-illness score for pediatric emergency patients. Pediatrics. 2005 Feb;115(2):388-95. doi: 10.1542/peds.2004-0586. PMID 15687449
- [Result] Lambert V, Matthews A, MacDonell R, Fitzsimons J. Paediatric early warning systems for detecting and responding to clinical deterioration in children: a systematic review. BMJ Open. 2017 Mar 13;7(3):e014497. doi: 10.1136/bmjopen-2016-014497. PMID 28289051
- [Result] Jagt EW. Improving Pediatric Survival from Resuscitation Events: The Role and Organization of Hospital-based Rapid Response Systems and Code Teams. Curr Pediatr Rev. 2013;9(2):158-74. doi: 10.2174/1573396311309020009. PMID 25417037
- [Result] Skaletzky SM, Raszynski A, Totapally BR. Validation of a modified pediatric early warning system score: a retrospective case-control study. Clin Pediatr (Phila). 2012 May;51(5):431-5. doi: 10.1177/0009922811430342. Epub 2011 Dec 8. PMID 22157421
- [Result] Egdell P, Finlay L, Pedley DK. The PAWS score: validation of an early warning scoring system for the initial assessment of children in the emergency department. Emerg Med J. 2008 Nov;25(11):745-9. doi: 10.1136/emj.2007.054965. PMID 18955610
- [Result] Barak-Corren Y, Fine AM, Reis BY. Early Prediction Model of Patient Hospitalization From the Pediatric Emergency Department. Pediatrics. 2017 May;139(5):e20162785. doi: 10.1542/peds.2016-2785. PMID 28557729